CLINICAL TRIAL: NCT00227929
Title: Effectiveness of Culturally Sensitive Collaborative Treatment (CSCT) of Depressed Chinese Americans in Primary Care
Brief Title: Culturally Sensitive Collaborative Treatment for Depressed Chinese Americans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Albert Yeung, Staff Psychiatrist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: K23MH067085 (NIH); K23MH067085 (NIH); DSIR 8K-RTSE
Record Dates: First submitted 2005-09-26; First posted 2005-09-28 (Estimated); Last update posted 2013-12-10 (Estimated); Status verified 2013-12

CONDITIONS: Depression
Keywords: Major Depressive Disorder; MDD
MeSH Terms: conditions — Depression; Depressive Disorder, Major

INTERVENTIONS:
Procedure: Care Management

SUMMARY:
This study will evaluate the effectiveness of culturally sensitive treatment versus regular care in treating depressed Chinese Americans.

DETAILED DESCRIPTION:
Depression is a complex illness that impacts an individual's thoughts, behavior, mood, and physical health. Research has shown that many Asian Americans with depression do not complain about their symptoms or seek treatment, which has lead to an under-recognition of depression in this population. Furthermore, even when a primary care physician does diagnose depression in an Asian American, adequate treatment does not often follow. There is a clear need to understand the cultural reasons for why treatment is not sought out by Asian Americans. There is also a need for developing new treatments that specifically target the Asian American population. Offering culturally sensitive therapies combined with traditional medical care may make depressed Asian Americans more comfortable in seeking treatment for their illness. Culturally Sensitive Collaborative Treatment (CSCT) is a comprehensive approach to treating depression. It incorporates consultation with a culturally trained psychiatrist, medical treatment provided by a primary care provider, and care management provided by a bilingual and bicultural care manager. The purpose of this study is to evaluate the effectiveness of CSCT versus traditional medical care for the treatment of depression in Chinese Americans.

This 24-week study will enroll depressed Chinese Americans. Potential participants will be interviewed in primary care clinics to screen for depression. Once enrolled, all participants will attend a consultation with a psychiatrist trained in cultural sensitivity to introduce the concept and treatment of depression. Participants will then be randomly assigned to either CSCT or standard care. Both groups of participants will receive regular care from their primary care provider, but the CSCT group will also meet with a bilingual and bicultural care manager to learn how to fully manage their depression. Outcome measurements will include symptoms of depression; adherence to appointments with primary care providers; adherence to medication treatment; and adverse events. All measurements will be assessed during follow-up phone calls at Weeks 2, 6, 10, 14, 18, 22, and 24.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity
* Currently depressed as determined by a total score of at least 16 on the CBCI scale
* Speaks and understands English or Chinese (including Mandarin, Cantonese, and Taiwanese dialect)
* Willing to participate in follow-up phone calls

Exclusion Criteria:

* Currently at risk for suicide
* Current unstable medical illness
* Current clinical or laboratory evidence of hypothyroidism
* Diagnosed with any of the following in addition to depression: organic mental disorder; schizophrenia; delusional disorder; psychotic disorder; bipolar disorder; mood congruent or mood incongruent psychotic features
* History of treatment by a psychiatrist within 4 months of study entry
* History of alcohol or substance abuse within 1 year of study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2003-07; Primary Completion 2007-09 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Symptoms of depression; measured at Weeks 2, 6, 10, 14, 18, 22, and 24

SECONDARY OUTCOMES:
Adherence to clinic visits with the primary care physicians; measured at Weeks 2, 6, 10, 14, 18, 22, and 24
Quality of life; measured at Weeks 2, 6, 10, 14, 18, 22, and 24
Adherence to medication treatment; measured at Weeks 2, 6, 10, 14, 18, 22, and 24
Adverse events; measured at Weeks 2, 6, 10, 14, 18, 22, and 24

CONTACTS AND LOCATIONS:
Overall Officials: Albert Yeung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- South Cove Community Health Center, Boston, Massachusetts, United States